CLINICAL TRIAL: NCT06908213
Title: Multicentric Evaluation of Enhanced Recovery After Surgery Protocol in Adolescent Idiopathic Scoliosis Surgery
Acronym: EMRACSIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL23_0742
Record Dates: First submitted 2025-03-07; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; adolescents; Enhanced recovery after surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, RIPH2
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : Improved Recovery After Surgery (Experimental): Patients in this group will undergo vertebral posterior fusion surgery with the Enhanced recovery after surgery protocol.
  This will include at least:
  * A one-day hospitalization to visit the surgical unit and to provide therapeutic education to patients and their parents.
  * A transition to morphine based treatments per os from intravenous morphine on the second day following surgery
  * Phone calls from a surgery unit nurse 2 times a day during 5 days
  * A teleconsultation with the surgeon between D3 and D5 following surgery Patients will also have a first consultation with the anesthesist and the surgeon then the surgery will be planned.
  They will also have 2 appointments at the hospital for post-surgical follow-up at D45 and M12.
  Interventions: Procedure: Posterior vertebral fusion surgery with Enhanced Recovery After Surgery (ERAS) procedure
- Control group (Experimental): Patients in this group will undergo posterior vertebral fusion surgery without the set of procedures for ERAS.
  They will have a first consultation with the anesthesist and the surgeon then the surgery will be planned. The discharge from hospital after surgery will not happen early and the standard of care procedures will be followed during and after surgery.
  Patients will receive 2 phone calls at D1 and D5 after surgery. The patient will also have 2 appointments at the hospital for post-surgical follow-up at D45 and M12.
  Interventions: Procedure: Posterior vertebral fusion surgery with standard of care procedure

INTERVENTIONS:
Procedure: Posterior vertebral fusion surgery with Enhanced Recovery After Surgery (ERAS) procedure — This will include at least:
  * A one-day hospitalization to visit the surgical unit and to provide therapeutic education to patients and their parents.
  * A transition to morphine based treatments per os from intravenous morphine on the second day following surgery
  * Phone calls from a surgery unit nurse 2 times a day during 5 days
  * A teleconsultation with the surgeon between D3 and D5 following surgery
  Arms: Experimental group : Improved Recovery After Surgery
Procedure: Posterior vertebral fusion surgery with standard of care procedure — Patients in this group will undergo posterior vertebral fusion surgery without the set of procedures for ERAS.
  They will have a first consultation with the anesthesist and the surgeon then the surgery will be planned. The discharge from hospital after surgery will not happen early and the standard of care procedures will be followed during and after surgery.
  Patients will receive 2 phone calls at D1 and D5 after surgery. The patient will also have 2 appointments at the hospital for post-surgical follow-up at D45 and M12.
  Arms: Control group

SUMMARY:
Adolescent idiopathic scoliosis is a deformation of the spine affecting 2 to 4% of under 18 years old population. This can have severe physical or psychological impact during adulthood. The deformation causes mechanical constraints resulting in early osteoarthritis, which results in adulthood disability.

There is also an impact on the respiratory function in most severe cases of idiopathic scoliosis. Adolescents affected by a scoliosis with an angle of 40° of more undergo a surgery called posterior fusion during adolescence to limit these impacts.

In France, more than 1000 adolescent patients undergo a surgery called posterior spinal fusion for their severe scoliosis.

This aims to straighten the spine by bone grafting all the vertebras included in the scoliosis. Two metal rods are implanted to favour osteosynthesis of the straight spine.

This intervention suffer of a bad image and worries the patients and their parents, as it needs metal implants near the spinal cord.

The worry comes from the most severe complication that may happen exceptionally following this surgery, which is a definitive paraplegia. The scar is quite large and the surgery reduces the mobility of a part of the spine. The intervention produces a quite large haemorrhage, which leads to a diminution in haemoglobin level, resulting in a fatigue during the following weeks.

On the following days, the patient will need a specific protocol of pain management including morphine-based and anti-inflammatory drugs.

This intervention will often require a 5 to 7 days hospitalization with a 1 to 2 month convalescence period at home or in rehabilitation centre.

This intervention is performed on adolescent patients without comorbidities. Moreover, the surgical approach is not profound passing between the para-vertebral muscles with no close large blood vessels or major organs. The pain is caused by correction tensions and the access to the vertebras during the surgery.

Surgical techniques have considerably evolved allowing shorter interventions and to reduce the loss of blood.

The association between morphine-based treatments and grade I analgesics enables an effective pain management.

This intervention appears to perfectly suit to an enhanced recovery after surgery procedure (ERAS).

ERAS is a set of procedure meant to enhance its tolerance and to reduce its morbidity and the hospitalization duration after surgery and the recovery duration.

ERAS is well developed in adult patients undergoing surgery, it is also well described in paediatric patient especially on adolescent scoliosis surgeries.

As the pain is well controlled during the hospitalization as well when the patient get back home, there are very few obstacles to an ERAS procedure in this indication for a patient without comorbidities.

Numerous articles report experiences of medical staff with ERAS protocols.

Generally, the set of measures includes:

* Before surgery: Providing information and therapeutic patient education, iron supplementation, physiotherapy, skin disinfection, digestive preparation against constipation
* During surgery: recuperations of blood cells to limit blood loss, use of modern tools to facilitate the positioning of pedicle screws, surgery performed by 2 surgeons
* After surgery: Pain management until stopping of analgesics by patient and maintenance of a link between the patient at home and the hospital staff after end of hospitalization The articles published about ERAS reports a favourable experience of such protocols with an efficient pain management, reduced hospitalization durations without increasing morbidity or re-hospitalizations. However, no studies have studied and proved by a robust scientific method the benefits of ERAS in adolescent scoliosis.

No studies evaluate the patients' quality of life or follow the patient for more than 6 months after surgery (limiting the assessment of long term complications e.g. infectious complications).

The link between hospital staff and the patient after his return back home is not described as well.

This research project aims to confirm with a robust scientific approach that ERAS protocols in idiopathic scoliosis in adolescents allow to reduce the duration of hospitalization compared to standard of care procedures while improving quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 11 and 17 years old
* Adolescent idiopathic scoliosis diagnosis
* Posterior vertebral fusion surgery indicated to treat the patient
* Informed consent signed by both parents / legal guardians

Exclusion Criteria:

* Comorbidities that might influence the duration of hospitalization (e.g. respiratory failure, diabetes…)
* Previous spine surgery
* Patient not benefiting from an health insurance plan
* Pregnant, parturient or breastfeeding woman
* Patient benefiting of psychiatric care
* Patient subject to a legal protection measure (guardianship, curatorship)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that ERAS in adolescent idiopathic scoliosis compared to standard of care procedure | At Month 3 (Collected on the day of discharge from surgery hospitalization)
  Hospitalization duration measured in days

SECONDARY OUTCOMES:
Improvement of quality of life at one day after return at home | Day 1 (VT1) after discharge from surgery hospitalization
  Quality of life questionnaires (PedsQL) at day 1 after return at home 4-point scale : 0 if it's never a problem
  1. if it's almost never a problem
  2. if it's sometimes a problem
  3. if it's often a problem
  4. if it's almost always a problem
Improvement of quality of life at 5 days, 45 days and 12 months after return at home | Day 1 (VT1), day 45 (V4) and month 12 (V5) after discharge from surgery hospitalization
  Quality of life questionnaires (PedsQL) at day 5, day 45 and month 12 after return at home 4-point scale : 0 if it's never a problem
  1. if it's almost never a problem
  2. if it's sometimes a problem
  3. if it's often a problem
  4. if it's almost always a problem
Changing post-surgical pain during hospitalization | Day 0 (V3), day 1 (VT1), day 5 (VT3); day 45 (V4) and month 12 (V5) after discharge from surgery hospitalization]
  Visual analog pain scale during surgery hospitalization 10-point scale: 0: no pain 10: uncontrollable pain
Changing post-surgical pain at day 1, day 5, day 45 and month 12 after return at home | Day 1 (VT1), day 5 (VT1), day 45 (V4) and month 12 (V5) after discharge from surgery hospitalization
  Visual analog pain scale 10-point scale: 0: no pain 10: uncontrollable pain
Changing post-surgical complications at day 45 and month 12 | Day 45 (V4) and month 12 (V5)
  Complications after surgery at day 45 and month 12 10-point scale: 0: no pain 10: uncontrollable pain
Changing the rate of re-hospitalization during the 12 months following surgery | From day of surgery day 0 (V3) to month 12 (V5)
  Re-hospitalization rate during the 12 monts following surgery
Describe the acceptability of the early discharge date from hospitalization in the two arms by patients and their parents | Day of surgery day 0 (V3)
  Percentage of parents refusal for early discharge date

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Amiens Site Sud, Amiens
  - CHU de Besançon Hopital Jean Minjoz, Besançon
  - Pediatric orthopedic surgery unit Hôpital femme Mère Enfant (HFME), Bron
  - CHU de Grenoble Hôpital Couple Enfant, La Tronche
  - Centre Medico-Chirurgical de Réadaptation des Massues Croix-Rouge, Lyon
  - AP-HM Hôpital de la Timone, Marseille
  - Fondation LENVAL, Nice
  - CHU de Saint-Etienne Hôpital Nord, Saint-Priest-en-Jarez
  - CHU de Toulouse, Toulouse
  - Clinique Médipôle Garonne, Toulouse
  - Clinique St Leonard, Trélazé

IPD SHARING:
Plan to Share IPD: No